CLINICAL TRIAL: NCT04062630
Title: Sacroiliac Joint Stabilization in Long Fusion to the Pelvis: Randomized Controlled Trial
Brief Title: SI Joint Stabilization in Long Fusion to the Pelvis
Acronym: SILVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300726
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Sacroiliac Joint Disruption; Scoliosis Lumbar Region
Keywords: Adult Scoliotic Spinal Deformity; Sacroiliac joint pain; multilevel lumbar surgery; SI Joint pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator): Multilevel Lumbar Fusion Surgery
  Interventions: Procedure: Multilevel Lumbar Fusion surgery
- Standard Care + iFuse 3-D (Experimental): Multilevel Lumbar Fusion Surgery with additional placement of iFuse 3-D in a trajectory parallel to the S2AI screws
  Interventions: Device: iFuse 3-D in Bedrock Configuration; Procedure: Multilevel Lumbar Fusion surgery

INTERVENTIONS:
Device: iFuse 3-D in Bedrock Configuration — Procedure in which 3 or more spinal segments are fused and concomitant pelvic fixation is performed, additionally iFuse 3-D implants are placed in a trajectory parallel to the S2AI screws.
  Arms: Standard Care + iFuse 3-D
Procedure: Multilevel Lumbar Fusion surgery — Procedure in which 3 or more spinal segments are fused and concomitant pelvic fixation is performed.

SUMMARY:
The purpose of this study is to compare outcomes of subjects undergoing multilevel lumbar fusion (MLF) surgery with and without the iFuse 3-D implants in the "bedrock" trajectory.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled, postmarket clinical study to determine the differences between subjects undergoing standard MLF surgery with S2AI fixation in the pelvis vs the additional placement of iFuse 3-D in the bedrock configuration during MLF surgery. Subjects will be monitored for sacroiliac (SI) joint pain and at two years post surgery a CT scan will be taken to assess S2AI screw loosening or any other findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-75 at time of screening
2. Patient scheduled for multilevel (>3 levels) spinal fusion surgery with planned fixation to the pelvis using S2AI screws
3. Patient has signed study-specific informed consent form
4. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements

Exclusion Criteria:

1. Indication for multilevel spine fusion surgery is any of the following:

   1. Congenital neuromuscular disease
   2. Prior pelvic fixation (i.e., patient already has S2AI or iliac bolts in place, current surgery indicated to revise this hardware)
   3. Grade IV spondylolisthesis
2. Prior sacroiliac joint fusion/fixation on either side
3. Presence of spinal cord stimulator
4. Presence of severe hip pain that could impair functional and quality of life improvement from complex spine surgery
5. Surgeon plans to use iliac screw for pelvic fixation
6. Any known sacral or iliac pathology
7. Any condition or anatomy that makes treatment with the iFuse Implant System infeasible
8. Known metabolic bone disease
9. Severe osteoporosis
10. Known allergy to titanium or titanium alloys
11. Use of medications known to have detrimental effects on bone quality and soft-tissue healing
12. Neurologic condition that would interfere with postoperative physical therapy
13. Current local or systemic infection that raises the risk of surgery
14. Patient currently receiving or seeking short- or long-term worker's compensation and/or currently involved in injury litigation related to the SI joint or low back pain.
15. Currently pregnant or planning pregnancy in the next 2 years
16. Prisoner or a ward of the state.
17. Known or suspected drug or alcohol abuse
18. Uncontrolled psychiatric disease that could interfere with study participation
19. Fibromyalgia

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion with S2AI screw abnormality on CT scan | 2 years
  Proportion of subjects with any of following: S2AI screw breakage, loosening or pullout OR rod breakage distal to S1 on 2-year CT scan as interpreted by an independent bone radiologist
Incidence of SI Joint pain | 2 years
  Proportion of subjects without SI joint pain at baseline who develop new onset SI joint pain by 2 years
Change from baseline in self-reported SI joint pain at 2 years | 2 years
  Change from baseline in self-reported SI joint pain on a 0 (no pain) -10 (worst imaginable pain) visual analog scale

SECONDARY OUTCOMES:
Proportion of subjects requiring revision, removal, reoperation or supplemental fixation | 2 years
  Proportion of subjects requiring revision, removal, reoperation or supplemental fixation related to S2AI screws or iFuse-3D
Therapeutic injection or other non-medication based intervention | 2 years
  Proportion of subjects requiring therapeutic injection or other non-medication based intervention to treat SI joint pain
Oswestry Disability Index | 2 years
  Change from baseline in self reported Oswestry Disability Index (ODI) score at 2 years
EuroQol Group Health Questionnaire | 2 years
  Change from baseline in self reported EuroQol Group Health Questionnaire with Time Trade Off Utility Index (EQ-5D TTO index) score at 2 years
Scoliosis Research Society 22r Patient Questionnaire | 2 years
  Change from baseline in self reported Scoliosis Research Society 22r Patient Questionnaire (SRS-22R) score at 2 years
Ambulatory and Work Status | 2 years
  Change from baseline in self reported ambulatory and work status at 2 years
Opioid Medication Use | 2 years
  Change from baseline opioid medications used, i.e., the mean daily dose during 2 weeks prior to each visit
Proportion of S2AI screw breakage | 2 years
  Proportion of S2AI screws with any breakage over the course of the study on CT scan as interpreted by an independent bone radiologist
Proportion of S2AI screw loosening | 2 years
  Proportion of S2AI screws with any loosening over the course of the study on CT scan as interpreted by an independent bone radiologist
iFuse-3D implant fully seated | 2 years
  Proportion of iFuse-3D implants placed fully seated (at least 20mm) into the sacrum on 2-year CT scan as interpreted by an independent bone radiologist
iFuse-3D implant position | 2 years
  Proportion of iFuse-3D implants with malposition (distal end outside of ilium) on 2-year CT scan as interpreted by an independent bone radiologist
Proportion of abnormal bone reactions in the pelvis | 2 years
  Proportion of abnormal bone reactions in the pelvis at either the iFuse-3D implant or S2AI screw on 2-year CT scan as interpreted by an independent bone radiologist
Change from baseline thoracic kyphosis at 2 years | 2 years
  Change from baseline thoracic kyphosis on 2-year CT scan as interpreted by an independent bone radiologist
Change from baseline pelvic tilt at 2 years | 2 years
  Change from baseline pelvic tilt on 2-year CT scan as interpreted by an independent bone radiologist
Change from baseline pelvic incidence at 2 years | 2 years
  Change from baseline pelvic incidence on 2-year CT scan as interpreted by an independent bone radiologist

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cher, MD, Study Director — SI-BONE
Locations (31):
- United States (27):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Hospital, La Jolla, California
  - University of California, San Diego, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - St Mary's Medical Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Orlando Health Physician Neurosurgery Group, Orlando, Florida
  - Axis Spine Center, Coeur d'Alene, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Buffalo Neurosurgery, Buffalo, New York
  - Hospital for Special Surgery, New York, New York
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - Tennessee Orthopaedics Alliance, Nashville, Tennessee
  - Austin Spine, Austin, Texas
  - North Texas Neurosurgical and Spine Center, Fort Worth, Texas
  - Texas Back Institute, Plano, Texas
  - UVA Spine Center - Ortho, Charlottesville, Virginia
  - University of Virginia - Dept of Neurosurgery, Charlottesville, Virginia
  - Ortho Virginia Research Institute, Richmond, Virginia
  - Virginia Mason, Seattle, Washington
- Epworth HealthCare, Richmond, Victoria, Australia
- Klinikum Magdeburg, Magdeburg, Germany
- Ospedale Civile di Legnano- ASST Ovest Milanese, Legnano, Milan, Italy
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data through Yale Open Data Access. Interested researcher may submit analysis plans to Yale.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After 2-year data are complete.
Access Criteria: Interested researcher may submit analysis plans to Yale Open Data Access program
URL: https://yoda.yale.edu/

REFERENCES:
- [Derived] Polly DW Jr. The Sacroiliac Joint: A Current State-of-the-Art Review. JBJS Rev. 2024 Feb 5;12(2). doi: 10.2106/JBJS.RVW.23.00151. eCollection 2024 Feb 1. PMID 38315777